CLINICAL TRIAL: NCT05078970
Title: Advancing Suicide Intervention Strategies for Teens During High Risk Periods
Acronym: ASSIST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Molly Adrian, Associate Professor, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01MH123442 (NIH)
Record Dates: First submitted 2021-09-22; First posted 2021-10-15 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Suicide Attempts; Suicidal Ideation; Suicide and Self-harm; Suicide Threat
MeSH Terms: conditions — Suicide, Attempted; Suicidal Ideation; Suicide; Self-Injurious Behavior | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1:1 ratio to
  1. Safety Planning Intervention plus follow up,
  2. Collaborative Assessment and Management of Suicidality, or
  3. usual care
Who Masked: Outcomes Assessor
Masking Description: Assessors will be blind to treatment assignment. It is not possible for clinicians or families to be blind to treatment procedures in psychotherapy since orientation to the model of care is part of psychotherapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment As Usual (TAU) (Active Comparator): Participants in this group will be studied as they proceed through treatment in the acute care setting and follow the intervention plan laid out in the discharge summary, per usual protocols at each facility. In both settings, the elements of typical care include crisis prevention planning, which outlines potential triggers, skills to use, and people and places to call in crisis, as well as referral to ongoing behavioral health treatment. We will not alter usual care but track recommendations, contacts and care through questionnaires the family completes as well as medical record review in order to understand the impact of the experimental conditions in relation to typical services.
  Interventions: Behavioral: Treatment As Usual
- Safety Planning Intervention+ (SPI+) (Active Comparator): SPI is focused on how the risk of suicidal crisis waxes and wanes over time. At times of heightened risk, a pre-specified and individualized plan targets the internal warning signs that become the cue to use the safety plan. SPI+ strategies focus on patient's narrative of the suicidal crisis and identifying solutions that are antithetical to progressing in a suicidal crisis. The brief structured intervention is conducted in six key steps. Youth in this condition will be offered weekly follow-up, with a minimum of 4 sessions and a maximum of 8 sessions. The goal is to create a crisis response plan to reduce risk when suicidal crises emerge. With adolescents, SPI+ consists of an individual session to elicit crisis narrative and motivation to utilize the safety plan through psychoeducation and follows six steps to achieve the adolescent's goals and return to safety when suicidal urges are high.
  Interventions: Behavioral: Safety Planning Intervention+ (SPI+)
- Collaborative Assessment and Management of Suicidality (CAMS) (Active Comparator): CAMS strategies focus on collaborative deconstruction and treatment of the patient-defined drivers- the problems that make suicide compelling to the patient- and utilizes these problem-focused treatment sessions to treat the drivers as directly related to wish to die. Participants will be assigned to CAMS for a minimum of 4 sessions and a maximum of eight sessions. This time frame, based on initial data from our pilot work with adolescents and emerging adults (18-25), suggests that a subset of participants resolve their STB in six to eight sessions. CAMS is a clinical intervention designed to modify how clinicians engage, assess and plan treatment with suicidal patients.
  Interventions: Behavioral: Collaborative Assessment and Management of Suicidality (CAMS)

INTERVENTIONS:
Behavioral: Safety Planning Intervention+ (SPI+) — SPI is focused on how the risk of suicidal crisis waxes and wanes over time. At times of heightened risk, a pre-specified and individualized plan targets the internal warning signs that become the cue to use the safety plan. SPI+ strategies focus on patient's narrative of the suicidal crisis and identifying solutions that are antithetical to progressing in a suicidal crisis. The brief structured intervention is conducted in six key steps. Youth in this condition will be offered weekly follow-up, with a minimum of 4 sessions and a maximum of 8 sessions. The goal is to create a crisis response plan to reduce risk when suicidal crises emerge. With adolescents, SPI+ consists of an individual session to elicit crisis narrative and motivation to utilize the safety plan through psychoeducation and follows six steps to achieve the adolescent's goals and return to safety when suicidal urges are high.
  Arms: Safety Planning Intervention+ (SPI+)
Behavioral: Collaborative Assessment and Management of Suicidality (CAMS) — CAMS strategies focus on collaborative deconstruction and treatment of the patient-defined drivers- the problems that make suicide compelling to the patient- and utilizes these problem-focused treatment sessions to treat the drivers as directly related to wish to die. Participants will be assigned to CAMS for a minimum of 4 sessions and maximum of eight sessions. This time frame, based on initial data from our pilot work with adolescents and emerging adults (18-25), suggests that a subset of participants resolve their STB in six to eight sessions. CAMS is a clinical intervention designed to modify how clinicians engage, assess and plan treatment with suicidal patients.
  Arms: Collaborative Assessment and Management of Suicidality (CAMS)
Behavioral: Treatment As Usual — This assigned condition tracks the care received in typical circumstances.
  Other Names: Usual Care
  Arms: Treatment As Usual (TAU)

SUMMARY:
To inform the effective management of adolescent suicide risk by evaluating promising treatments and developing the evidence-base for interventions that are well suited for widespread adoption, sustained quality, and impact.

DETAILED DESCRIPTION:
The current study aims to evaluate Safety Planning Intervention with follow-up (SPI+), Collaborative Assessment and Management of Suicidality (CAMS) and usual care. Adolescents, parents, and clinicians will participate in the project to advance to following Research Aims: 1) Assess the comparative effectiveness of CAMS and SPI+ compared to usual care, 2) Evaluate the mechanism of change accounting for the therapeutic effects of the interventions 3) Identify moderators of treatment effects. Participants and their parents will receive study assessments at baseline, 2-week, 1-month, 2-month, 6-month, and 12-month timepoints. Study assessments will ask about participant demographics (sample characterization), suicide attempts, suicidal ideation, non-suicidal self-injury, service utilization, self-assessed risk, treatment integrity, sleep, family cohesion, and social experiences. Youth participants and their legal guardian both consent to participate in the research procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Youth, aged 11-17
3. Endorse suicidal ideation and/or behavior
4. Admitted to acute care (emergency, inpatient medical or inpatient psychiatric) due to suicidality

Exclusion Criteria:

1. Presence of psychosis, intellectual disability, autism spectrum disorder, eating disorder with unstable vitals
2. Limited English proficiency that would interfere with the ability to complete study assessments

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 306 (Estimated)
Dates: Start 2022-08-11 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Suicidal events | Suicidal events at 12 months
  Change the rate of suicidal events as measured by death by suicide, attempted suicide, preparatory acts toward imminent suicidal behavior, or suicidal ideation resulting in a change in treatment plan or emergency evaluation as measured by the C-SSRS.

SECONDARY OUTCOMES:
Suicide attempts | Suicide attempts at 12 months
  Self injurious behavior with intent to die as measured by the C-SSRS
Suicidal Ideation | Change in score from baseline to 12 months
  Severity of suicidal ideation as measured by the total score on the Suicidal Ideation Questionnaire Junior (SIQ-Jr. This 15 item measure is rated on a Likert scale, with scores ranging from 0 to 90, with higher scores reflecting worse outcomes and more severe ideation.

CONTACTS AND LOCATIONS:
Overall Officials: Molly Adrian, Principal Investigator — Seattle Childrens
Locations (2):
- United States (2):
  - Nationwide Children's, Columbus, Ohio
  - Seattle Children's, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Data will be submitted to the National Institute of Mental Health Data Repository
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available in the NIMH NDA 1 year from study completion.
Access Criteria: NIMH NDA access criteria applies.

REFERENCES:
- [Derived] Adrian M, McCauley E, Gallop R, Stevens J, Jobes DA, Crumlish J, Stanley B, Brown GK, Green KL, Hughes JL, Bridge JA. Advancing Suicide Intervention Strategies for Teens (ASSIST): study protocol for a multisite randomised controlled trial. BMJ Open. 2023 Dec 12;13(12):e074116. doi: 10.1136/bmjopen-2023-074116. PMID 38086585